CLINICAL TRIAL: NCT00045734
Title: Phase II Trial of STI571 (NSC 716051) in Patients With Recurrent Meningioma
Brief Title: Imatinib Mesylate in Treating Patients With Recurrent Meningioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02495; NABTC-0108; U01CA062399 (NIH); CDR0000257267 (Registry Identifier: PDQ (Physician Data Query)); NCT00069667 (obsolete NCT alias)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Adult Grade I Meningioma; Adult Grade II Meningioma; Adult Grade III Meningioma; Adult Meningeal Hemangiopericytoma; Adult Meningioma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Meningioma; Brain Neoplasms | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate once or twice daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Other: pharmacological study/ laboratory biomarker analysis
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase II trial to study the effectiveness of imatinib mesylate in treating patients who have recurrent meningioma. Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the efficacy of imatinib mesylate, in terms of 6-month progression-free survival, of patients with recurrent meningioma.

SECONDARY OBJECTIVES I. Determine the response rate and overall survival of patients treated with this drug.

II. Evaluate the safety profile of this drug in these patients. III. Determine the pharmacokinetics of this drug in these patients. IV. Develop exploratory data concerning surrogate markers of of angiogenic activity in vivo using functional neuro-imaging studies and in vitro assays of serum angiogenic peptides of this drug in these patients.

V. Develop exploratory data concerning evidence of platelet-derived growth factor (PDGF) inhibition in tumor specimens taken from patients undergoing surgery VI. Develop exploratory data correlating molecular abnormalities in the tumor with response in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to concurrent use of enzyme-inducing antiepileptic drugs (yes vs no), histology (benign vs atypical or malignant), neurofibromatosis positivity (yes vs no), and preoperative candidacy (yes vs no).

Patients receive oral imatinib mesylate once or twice daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 60 patients (30 per stratum) will be accrued for this study within 8-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed meningioma

  * Benign, malignant, or atypical disease
  * Neurofibromatosis (NF) type 1 or 2 allowed
  * Hemangiopericytoma allowed
* Unequivocal evidence of tumor recurrence or progression by MRI or CT scan (on steroid dosage that is stable for at least 5 days)
* Evaluable residual disease by MRI or CT scan if previously treated with surgical resection for recurrent or progressive disease
* Newly diagnosed recurrent disease that requires surgical debulking allowed
* Prior standard external-beam radiotherapy, interstitial brachytherapy, or gamma-knife radiosurgery allowed provided disease has progressed since completion of therapy

  * Patients who have had prior brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based upon positron-emission tomography or thallium scanning, magnetic resonance spectroscopy, or surgical documentation
* Patients with a history of NF may have other stable Central Nervous System (CNS) tumors (e.g., schwannoma, acoustic neuroma, or ependymoma) provided those lesions have been stable in size for the past 6 months
* Performance status - Karnofsky 60-100%
* More than 8 weeks
* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 120,000/mm^3
* Hemoglobin at least 10 g/dL (transfusions allowed)
* No bleeding disorders
* Bilirubin less than 2 times upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) less than 2 times ULN
* Prothrombin Time (PT), Partial thromboplastin time (PTT), and International normalized Ratio (INR) no greater than 1.5 times ULN
* Creatinine less than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No deep venous or arterial thrombosis within the past 6 weeks
* No pulmonary embolism within the past 6 weeks
* No serious active infection
* No prior intracranial hemorrhage
* No concurrent disease that would obscure toxicity or dangerously alter drug metabolism
* No other malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix unless the patient is in complete remission and off all therapy for that disease for at least 3 years
* No other significant medical illness that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study participation
* At least 1 week since prior interferon or thalidomide
* No concurrent immunotherapy
* Concurrent epoetin alfa allowed
* At least 4 weeks since prior cytotoxic chemotherapy
* At least 2 weeks since prior vincristine
* At least 6 weeks since prior nitrosoureas
* At least 3 weeks since prior hydroxyurea or procarbazine
* No concurrent chemotherapy
* At least 1 week since prior tamoxifen
* No concurrent hormonal therapy
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy
* Recovered from prior surgery
* Recovered from all prior therapy
* At least 1 week since prior noncytotoxic therapy (e.g., isotretinoin) except radiosensitizers
* At least 2 weeks since prior drugs that affect hepatic metabolism
* At least 4 weeks since prior investigational agents
* No concurrent warfarin (heparin or low-molecular weight heparin allowed)
* No other concurrent investigational agents
* No concurrent acetaminophen of more than 500 mg/day
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wen, MD, Principal Investigator — North American Brain Tumor Consortium
Locations (7):
- United States (7):
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - National Cancer Institute Neuro-Oncology Branch, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients enrolled between June 2003 ad August 2005 in an outpatient clinic setting.
Groups:
- Treatment (Imatinib Mesylate): Patients receive oral imatinib mesylate once or twice daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Other: pharmacological study/ laboratory biomarker analysis
  imatinib mesylate: Given orally
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Imatinib Mesylate)
Started | 23
Completed | 22
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: 23 patients were enrolled and evaluated however 1 patient was found to be ineligible as patient had a second malignancy within 3 years of registration. Demographics for this patient are reported.
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 58 [26 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Karnofsky Performance Status Scale (KPS) [Median (Full Range); unit: units on a scale] — High best 100 normal no complaints no disease 90 capable of normal activity few symptoms/disease 80 normal activity w/ some difficulty some symptoms/signs 70 caring for self not capable of normal activity/work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care/help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures/treatment 10 moribund rapidly progressive fatal disease processes 0 death
  units on a scale | 80 [60 to 100]
Histology [Number; unit: participants] — using the WHO classification histology code which is the International classification for Oncology
  Benign (WHO grade I) Atypical (WHO grade II) Anaplastic (WHO grade III)
  participants
    Benign (WHO grade I) | 13
    Atypical (WHO grade II) | 5
    Anaplastic (WHO grade III) | 5
Prior Surgeries [Median (Full Range); unit: surgeries] | 3 [1 to 8]
Prior Radiation Therapies [Median (Full Range); unit: Radiation Therapies] | 1 [0 to 5]
Prior Chemotherapy Regimens [Median (Full Range); unit: Chemotherapy Regimens] | 0 [0 to 2]

OUTCOME MEASURES:

1. Primary Outcome: 6 Months - Progression-free Survival According to Response Evaluation Using Macdonald Criteria
Description: The Macdonald criteria, roughly similarly to other systems, divides response into 4 types of response based on imaging (magnetic resonance imaging [MRI]) and clinical features
  1: complete response; 2: partial response; 3:stable disease; 4:progression
  Complete response imaging features: disappearance of all enhancing disease (measurable and non-measurable) sustained for at least 4 weeks; no new lesions clinical features; no corticosteroids; clinically stable or improved
  Partial response imaging features: 50% or more decrease of all measurable enhancing lesions sustained for at least 4 weeks: no new lesions clinical features: stable or reduced corticosteroids; clinically stable or improved
  Stable disease imaging features: does not qualify for complete response, partial response or progression clinical features: clinically stable
  Progression imaging features: 25% of more increase in enhancing lesions; any new lesions clinical features: clinical deterioration
Time Frame: At 6 months
Population: Only 19 of the 23 patients were evaluable for response
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 19
percentage of participants | 29.4

2. Secondary Outcome: Progression-free Survival According to Response Evaluation Using Macdonald Criteria
Description: The Macdonald criteria, roughly similarly to other systems, divides response into 4 types of response based on imaging (MRI) and clinical features
  1: complete response; 2: partial response; 3:stable disease; 4:progression
  Complete response imaging features: disappearance of all enhancing disease (measurable and non-measurable) sustained for at least 4 weeks; no new lesions clinical features; no corticosteroids; clinically stable or improved
  Partial response imaging features: 50% or more decrease of all measurable enhancing lesions sustained for at least 4 weeks: no new lesions clinical features: stable or reduced corticosteroids; clinically stable or improved
  Stable disease imaging features: does not qualify for complete response, partial response or progression clinical features: clinically stable
  Progression imaging features: 25% of more increase in enhancing lesions; any new lesions clinical features: clinical deterioration
Time Frame: 3 years
Population: Of the 22 eligible patients only 19 were evaluable for response
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 19
months | 2 [0.7 to 34]

3. Secondary Outcome: Toxicity as Assessed by the Cancer Therapy Evaluation Program Common Toxicity Criteria (CTC) Version 2.0
Description: percentage of patients who had grade 3 or grade 4 adverse events
Time Frame: Up to 5 years after completion of study treatment
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 23
percentage of patients | 2.3

4. Secondary Outcome: Tumor Response as Assessed by MRI Using Macdonald Criteria
Description: as for outcome 2
Time Frame: Up to 5 years
Population: response at first scan
Measure: Number; unit: participants
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 19
participants
  Progression | 10
  Stable | 9

5. Secondary Outcome: Concentration (Steady State) of Imatinib During Cycle One (Pharmacokinetics)
Description: Blood collected before and at 1,2,4 ad 24 hours after ingestion of imatinib on day 8 of cycle 1
  result is the measurement of the before dosing on day 8 (trough level) and the 24 hour dosing day 8
Time Frame: pre dosing on day 8 and 24 hour dosing day 8 of Pre-dosing Day 9
Population: Only 14 samples available / evaluable for analysis
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 22
ng/ml
  Day 8 Pre Dosing: number analyzed (Participants) | 14
  Day 8 Pre Dosing | 2129 (1600)
  Day 8 24 hour dosing: number analyzed (Participants) | 14
  Day 8 24 hour dosing | 2248 (1408)

6. Secondary Outcome: Determine Survival for Patients Treated With Imatinib Mesylate
Description: survival determined from start of treatment to date of death
Time Frame: 3 years
Population: death date of 7 patients were unknown at time of analysis
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 17
months | 16.8 [2.1 to 48.6]

7. Other Pre Specified Outcome: Determine Surrogate Markers of Angiogenic Peptides Using Functional Neuro-imaging and in Vitro Bioassays
Description: Study terminated early, only 22 patients entered on study. Hence, this secondary outcome was never analyzed due number of patients.
Time Frame: 5 years
Population: Study terminated early, only 22 patients entered on study. Hence, this secondary outcome was never analyzed due to number of patients.
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Evidence of Platelet-derived Growth Factor (PDGF) Inhibition in Tumor Specimens
Description: insufficient samples to allow Platelet-derived growth factor receptor (PDGFR-alpha and -beta expression to be correlated Of 22 patients only 7 samples available and only 5 yielded adequate tissue
Time Frame: - 3 years
Population: insufficient samples to allow PDGFR-alpha and -beta expression to be correlated Of 22 patients only 7 samples available and only 5 yielded adequate tissue
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Determine Correlating Molecular Abnormalities in the Tumor With Response to Treatment
Description: Measurable: Bidimensionally measurable lesions w/ clearly defined margins by MRI Evaluable: Unidimensionally measurable lesions, masses w/margins not clearly defined.
  Complete Response (CR): Complete disappearance of all measurable/evaluable disease. No new lesions. No evidence of non-evaluable disease. Patients on minimal/no steroids.
  Partial Response (PR): >/= to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. Responders must be on same/decreasing doses of dexamethasone.
  Stable/No Response: Does not qualify for CR, PR, or progression. Progression: 25% increase in the sum of products of all measurable lesions over smallest sum observed (over Baseline (BL) if no decrease), OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 3 years
Population: as for outcome 7
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Treatment (Imatinib Mesylate)
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 10/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Imatinib Mesylate) (N=22)
anemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
CNS (intracranial) Hemorrhage (Nervous system disorders) | 1 (1)
dehydrations (Metabolism and nutrition disorders) | 1 (1)
dizziness (Nervous system disorders) | 1 (1)
elevated serum glutamic pyruvic transaminase (Investigations) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was closed prematurely due to limited activity and slow accrual. Study was designed to enroll (statistically powered) for 30 patients into each group (30 benign; 30 Atypical and 30 Anaplastic) meningioma's. Study enroll only 23 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less